CLINICAL TRIAL: NCT06318832
Title: Optimizing a Wellbeing Program for Care-partners of Those With Spinal Cord Injury
Brief Title: Optimizing a Wellbeing Program for Care-partners of Those With SCI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Swati Mehta, Scientist, Principle Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 124609
Record Dates: First submitted 2024-03-13; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Internet-Delivered Cognitive Behavioural Therapy; Depression; Anxiety; Spinal Cord Injuries; Caregiver Burnout
MeSH Terms: conditions — Depression; Anxiety Disorders; Spinal Cord Injuries; Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Internet Delivered Cognitive Behavioural Therapy (ICBT) (Experimental): ICBT: Participants will receive the 10-week tailored ICBT Wellbeing program consisting of 1) education about how taking on the role of care-partner can impact emotional and cognitive wellbeing through introduction to the CBT model; 2) structured problem solving; 3) cognitive therapy and thought challenging to manage one's wellbeing and impact of caregiving; 4) building communication and intimacy; 5) physical symptoms of depression (i.e., hypo-arousal), anxiety/anger (i.e., hyper-arousal); practicing behavioural activation and controlled relaxation; 6) overdoing-underdoing cycle of activity levels and issues around the fear avoidance of social, physical, and cognitive activities; practicing activity pacing and gradually tackling avoidance; 7) occurrence of setbacks in thought, physical, behavioural, and cognitive symptoms; signs of setbacks and creating setback plans.
  Interventions: Other: ICBT
- ICBT and Therapist Guidance (TG) (Active Comparator): ICBT Therapist Guidance: Weekly Guidance will be provided by a Guide who is a registered social worker with a Master's in Social Work. The Guide will spend ~15 -20 mins. per week/per participant. Weekly interaction will consist of: 1) assist participants practice skills, reinforce progress, engage with the program; 2) guide participants to learn material, highlight lesson content, answer questions, and problem solve on how to apply skills; 3) provide support through warmth and concern; 4) monitor symptoms and risk management.
  Interventions: Other: ICBT
- ICBT and Peer Support (PS) (Active Comparator): ICBT Focused Peer Group Discussion: The focused discussion will take the form of a group based virtual session of approximately 6-8 participants in each group The Groups will be moderated by a Spinal Cord Injury Ontario Client Services team member once every two weeks for the duration of the 10-week program.
  Interventions: Other: ICBT
- ICBT and Booster (B) (Active Comparator): ICBT
  Booster sessions: Participants allocated to receive booster sessions will have access to a booster module at 16 weeks post enrollment. The booster module will include online materials that review core skills such as thought challenging, deep breathing, behavioural activation, and graded exposure. The module will also discuss how to maintain motivation and continue to practice skills regularly. The Booster module will also include a Do-It-Yourself Guide for participants to print and practice the skills they have learned throughout the course.
  Interventions: Other: ICBT
- ICBT+TG+PS (Active Comparator): ICBT and TG and PS
  Interventions: Other: ICBT
- ICBT+TG+B (Active Comparator): ICBT and TG and B
  Interventions: Other: ICBT
- ICBT+PS+B (Active Comparator): ICBT and PS and B
  Interventions: Other: ICBT
- ICT+TG+PS+B (Active Comparator): ICBT and TG and PS and B
  Interventions: Other: ICBT

INTERVENTIONS:
Other: ICBT — ICBT: Participants will receive the 10-week tailored ICBT Wellbeing program consists of 1) education about how taking on the role of care-partner can impact emotional and cognitive wellbeing through introduction to the CBT model; 2) structured problem solving; 3) cognitive therapy and thought challenging to manage one's wellbeing and impact of caregiving; 4) building communication and intimacy; 5) physical symptoms of depression (i.e., hypo-arousal), anxiety/anger (i.e., hyper-arousal); practicing behavioural activation and controlled relaxation; 6) overdoing-underdoing cycle of activity levels and issues around the fear avoidance of social, physical, and cognitive activities; practicing activity pacing and gradually tackling avoidance; 7) occurrence of setbacks in thought, physical, behavioural, and cognitive symptoms; signs of setbacks and creating setback plans.

SUMMARY:
Spinal cord injuries (SCI) have a devastating effect not only on individuals incurring the life changing event, but also on those who are involved in their care. Family care-partners of those with SCI (fcSCI) may experience significant negative effects including impaired mental health, high levels of burden, poor adjustment to role, decreased quality of life and strain on relationships. Cognitive behaviour therapy (CBT) is an evidence-based treatment strategy that helps individuals recognize and challenge their unhelpful thoughts and behaviours that contribute to their mental health concerns. However, barriers such as availability to specialized care, costs, rural and remote location, or concerns about stigma may limit access to care. Internet delivered CBT (ICBT) has the potential to reach a much wider group of people that may have unequal access to health care.

In a previous feasibility study, the team demonstrated the preliminary effectiveness of a tailored ICBT Wellbeing program for fcSCI. However, our understanding of which components of the program can result in optimal management is limited. The main purpose of this study is to evaluate the effectiveness of different components of the Wellbeing program including: therapist guidance, peer support groups, and booster sessions on symptoms of depression among fcSCI. The team will evaluate which intervention components result in meaningful improvement in symptoms of depression. Through collaborations with SCI community organizations and rehabilitation institutions, participants will be recruited across Canada. The researchers will also develop a model to examine the most cost-effective intervention package from the different components. The Wellbeing for fcSCI program can provide personalized service to individuals while being flexible and easily accessible, improving overall wellbeing and access to health care services.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Canadian residents
3. identify as fcSCI
4. living in the community
5. endorsing symptoms of depression (PHQ-9≥5);
6. suicide risk score <8 (Suicide Behaviours Questionnaire (SBQ) (Osman et al. 2001)
7. speak and read English
8. able to access and be comfortable using computers and the internet
9. willing to provide the name of a physician as an emergency contact.

Exclusion Criteria:

1. are currently involved in another psychotherapeutic intervention
2. present with severe mental health disorder requiring face-to-face therapy (e.g., severe suicide ideation, severe substance abuse, recent history of psychosis, mania).

Those participants taking antidepressants will be included in the trial; medication use will be tracked.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Change in depression | Baseline to 1 year follow up
  Patient Health Questionnaire - 9 Item (PHQ-9). Higher total scores indicate greater severity of depression. Scores range from 0 to 27.